CLINICAL TRIAL: NCT00781794
Title: A Double-Blind, Placebo-Controlled, Crossover Study to Evaluate the Effects of Single Oral Doses of NSA-789 on Auditory P50 Suppression in Nonsmoking Patients With Stabilized Schizophrenia
Brief Title: Study Evaluating The Effects Of Single Oral Doses Of NSA-789 On Auditory P50 Suppression In Schizophrenic Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 3230A1-1005
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Dose 1
  Interventions: Drug: NSA-789 at 2 different doses
- 2 (Experimental): Dose 2
  Interventions: Drug: NSA-789 at 2 different doses
- 3 (Placebo Comparator)
  Interventions: Drug: NSA-789 at 2 different doses

INTERVENTIONS:
Drug: NSA-789 at 2 different doses

SUMMARY:
The purpose of this study is to evaluate the effect of single doses of NSA-789 on the P50 component of the auditory evoked potentials and to assess the safety, tolerability and the concentration of NSA-789 in the blood, in nonsmoking patients with schizophrenia.

ELIGIBILITY:
Inclusion criteria:

* Women of nonchildbearing potential, or men, aged 18 to 55 years inclusive on study day 1. Women of nonchildbearing potential may be included if they are either surgically sterile (hysterectomy and/or oophorectomy) or postmenopausal for â‰¥1 year (with a follicle-stimulating hormone [FSH] level of â‰¥38 mIU/mL). Women who are surgically sterile must provide documentation of the procedure by an operative report or ultrasound scan. Sexually active men must agree to use a medically acceptable form of contraception during the study and continue it for 12 weeks after test article administration.
* Body mass index in the range of 18 to 32 kg/m2 and body weight â‰¥50 kg.
* Hemoglobin no lower than 0.4 g/dL, less than the lower limit of the normal range, and white blood cell count no lower than 0.5 103/mm3, less than the lower limit of the of the normal range at screening and day -1. Hematocrit and absolute neutrophil count within normal range at screening and on day -1.

Exclusion criteria:

* Women of childbearing potential.
* Presence or history of any disorder that may prevent the successful completion of the study.
* Any unstable psychiatric condition, which may prevent the successful and safe completion of the study in the opinion of the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01 (Estimated); Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
electroencephalogram | 8 weeks

SECONDARY OUTCOMES:
blood sample | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (3):
- Glendale, California, United States
- France (2):
  - Rouffach
  - Toul